CLINICAL TRIAL: NCT05999721
Title: The Effect of Superficial Parasternal Intercostal Plane Block on Pulmonary Function Tests After Cardiac Surgery (PIPACS Trial): a Prospective, Double-blind, Randomised Controlled Trial.
Brief Title: The Effect of Superficial Parasternal Intercostal Plane Block on Pulmonary Function Tests After Cardiac Surgery
Acronym: PIPACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shai Fein (Other)
Responsible Party: Sponsor-Investigator, Shai Fein, Principal Investigator, Head of Department, Department of Anesthesia, Beilinson Hospital, Rabin Medical Centre, Petach Tikva, Israel., Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0577-23-RMC
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain; Pulmonary Function Tests
Keywords: Superficial Parasternal Intercostal Plane Block; Pulmonary function tests; Cardiac surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): In addition to standard care, the treatment arm will receive an ultrasound-guided bilateral single-shot superficial parasternal intercostal plane block at two levels.
  Interventions: Procedure: superficial parasternal intercostal plane block; Other: Standard care
- Control Arm (Active Comparator): The control arm will receive standard care alone.
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: superficial parasternal intercostal plane block — Injection of 60 mL of bupivacaine 0.25% and epinephrine 2.5 µg mL-1
  Arms: Treatment Arm
Other: Standard care — Operating Room:
  Anaesthesia will be induced using midazolam (0.1-0.15 mg kg-1), fentanyl (5-10 μg kg-1), and rocuronium (0.6-1.2 mg kg-1); then, after tracheal intubation, anaesthesia will be maintained using isoflurane at one MAC, along with continuous fentanyl (3-5 μg kg-1 h-1) and midazolam (20-50 μg kg-1 h-1). Additional boluses of fentanyl will be administered according to the anesthesiologist's discretion.
  Cardiothoracic Intensive Care Unit:
  Continuous fentanyl will be maintained until tracheal extubation. All patients will receive intravenous multimodal analgesic drugs around the clock, including paracetamol 3 g day-1 and dipyrone 3 g day-1. If pain persists, rescue doses of either intravenous tramadol or morphine will be administered.
  Cardiothoracic ward:
  The analgesic protocol includes around-the-clock intravenous paracetamol 3 g day-1 and dipyrone 3 g day-1. If pain continues, rescue doses of oral oxycodone will be administered.

SUMMARY:
In adult patients undergoing cardiac surgery, does adding an sPIP block to standard care compared to standard care alone result in a smaller decrease in PFTs?

DETAILED DESCRIPTION:
Postoperative pulmonary complications are a significant concern after cardiac surgery, with post-sternotomy pain contributing to impaired pulmonary function and increased risk of these complications. Parasternal intercostal plane blocks have recently emerged as a promising analgesic option for cardiac surgery, but their impact on pulmonary function tests (PFTs) has yet to be evaluated.

This prospective, single-center, double-blind, randomized controlled trial will recruit 100 adult patients undergoing elective cardiac surgery. Baseline pulmonary function, including FEV1, FVC, and PEF, will be measured preoperatively and reassessed on the first postoperative day to evaluate the primary outcome: percentage change in PFT values. Secondary outcomes include pain scores, opioid consumption, incidence of postoperative pulmonary complications during hospitalization, duration of cardiothoracic intensive care and hospital stays, and 30-day mortality.

This study aims to determine whether adding a superficial parasternal intercostal plane (sPIP) block to standard care better preserves pulmonary function in adult patients undergoing elective cardiac surgery.

ELIGIBILITY:
Inclusion criteria:

* Patients who are scheduled to undergo elective cardiac surgery via sternotomy (i.e., coronary artery bypass graft, valvular surgery, and combined surgery).
* Body Mass Index (BMI) above 20 and below 40 kg m-2
* Age above 18 years.
* Eligible to sign informed consent.

Exclusion criteria:

* Change from scheduled morning surgery to a non-morning case or emergency surgery.
* Redo surgery.
* Off-pump surgeries.
* Pregnancy.
* Preoperative mechanical circulatory support (i.e., intra-aortic balloon pump, extracorporeal membrane oxygenation, ventricular assist devices).
* Preoperative chronic pain (i.e., fibromyalgia, chronic neuropathic pain).
* Contraindication for regional analgesia (i.e., known allergy to LA, skin lesions in the injection site).
* Known allergy to one or more of the components of multimodal analgesia (i.e., opioids, paracetamol, tramadol, dipyrone).
* Preexisting severe pulmonary disease (i.e., an obstructive lung disease with FEV1 below 49%, restrictive lung disease with FVC below 49%, pulmonary hypertension).
* Patients requiring mechanical ventilation for more than 24 hours postoperatively.

Criteria For Discontinuing (Postoperative Exclusion Criteria):

* Prolonged cardiopulmonary bypass (CPB) of more than three hours.
* Transfusion of more than three units of blood products.
* Severe coagulation disturbance requiring prothrombin complex concentrate or recombinant factor VII.
* Left ventricular failure with vasoactive-inotropic score (VIS) at the end of the surgery of ≥ 20.
* Right ventricular failure requires inhaled nitric oxide.
* Need for mechanical circulatory support (i.e., intra-aortic balloon pump, extracorporeal membrane oxygenation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Forced Expiratory Volume in the First Second (FEV1) | Baseline (preoperative) and first postoperative day
  Percentage change in FEV1 (measured in litres) from baseline to the first postoperative day.
Percentage Change in Forced Vital Capacity (FVC) | Baseline (preoperative) and first postoperative day
  Percentage change in FVC (measured in litres) from baseline to the first postoperative day.
Percentage Change in Peak Expiratory Flow (PEF) | Baseline (preoperative) and first postoperative day
  Percentage change in PEF (measured in litres per second) from baseline to the first postoperative day.

SECONDARY OUTCOMES:
Pain scores, measured by Numeric Rating Scale (NRS) | 0-8 hours, 8-16 hours, 16-24 hours, 24-48 hours, and 48-72 hours postoperatively
  Maximum pain NRS (0-10) recorded at various time intervals.
Opioid consumption, measured in Morphine Milligram Equivalents (MME) | 0-8 hours, 8-16 hours, 16-24 hours, 24-48 hours, and 48-72 hours postoperatively
  Opioid consumption measured in MME at various time intervals postoperatively.
Postoperative pulmonary complication, based on the European perioperative clinical outcome (EPCO) criteria | 30 days
  The incidence of postoperative pulmonary complications during current hospitalisation
Length of stay | 30 days
  The length of cardiothoracic intensive care unit and hospital stay
Mortality | 30 days
  Thirty-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Shai Fein, MD, MHA, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No
Participant-level datasets and statistical code will be provided upon request.